CLINICAL TRIAL: NCT01886677
Title: Exploring the Impact of Negative Energy Balance in Men With Prostate Cancer
Brief Title: Improving Energy Balance in Men With Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Wendy Demark-Wahnefried, PhD, Professor and Webb Endowed Chair of Nutrition Sciences Associate Director, UAB Comprehensive Cancer Center, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R21CA161263-01A1 (NIH)
Record Dates: First submitted 2013-06-19; First posted 2013-06-26 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2014-12

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; intervention; diet; physical activity; exercise; weight loss; biomarkers; cancer progression
MeSH Terms: conditions — Prostatic Neoplasms; Motor Activity; Weight Loss; Disease Progression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate diet and exercise intervention (Experimental): A healthful diet plus exercise intervention to promote a weight loss of up to 2 pounds/week
  Interventions: Behavioral: Immediate diet and exercise intervention
- Delayed diet and exercise intervention (Other): This arm will receive the same diet and exercise intervention as the experimental arm once recovery from prostatectomy is achieved.
  Interventions: Behavioral: Delayed diet and exercise intervention

INTERVENTIONS:
Behavioral: Immediate diet and exercise intervention — Both arms will receive the same intervention: a healthful diet plus exercise intervention to promote a weight loss of up to 2 pounds/week. The only difference is the timing of the delivery of the intervention (immediate vs. delayed).
  Arms: Immediate diet and exercise intervention
Behavioral: Delayed diet and exercise intervention — Both arms will receive the same intervention: a healthful diet plus exercise intervention to promote a weight loss of up to 2 pounds/week. The only difference is the timing of the delivery of the intervention (immediate vs. delayed).
  Arms: Delayed diet and exercise intervention

SUMMARY:
RATIONALE: Obesity and overweight are associated with the risk of aggressive disease, and energy balance may play a major role in prostate cancer progression.

PURPOSE: Randomized phase II trial to study the effectiveness of weight loss, via a healthy energy-restricted diet and exercise, in slowing or preventing disease progression in patients who have newly diagnosed prostate cancer.

DETAILED DESCRIPTION:
This is a 2-arm randomized controlled feasibility trial among 40 overweight or obese men newly diagnosed with prostate cancer who are scheduled for prostatectomy. This study will use the presurgical period to explore the potential impact of weight loss via a healthy energy-restricted diet and increased physical activity on circulating hormones, cytokines, and growth factors, as well as effects on tumor biology and other clinical outcomes. Consenting patients will be block randomized to 1-of-2 study arms: 1) a healthful diet + exercise intervention to promote a weight loss of up to 2 pounds/week; or 2) a wait-list control who will receive the intervention once the study period is complete. Both groups will receive nutritional counseling during the study period to correct nutritional deficiencies with food sources. This study will explore and contrast changes in body mass index (BMI) observed over the study period (minimum of 3.5 weeks) in the intervention vs. wait-list control arms, and also monitor changes in body composition, energy intake and physical activity; these changes will be studied in relation to the following endpoints: a) changes in select circulating biomarkers and gene expression related to cancer progression, hormonal status, inflammation and other energy-related factors; b) rates of tumor proliferation and apoptosis; c) tumor immunohistochemical markers of insulin receptor, vascular endothelial growth factor (VEGF), AKT, and nuclear factor kappa-light-chain-enhancer of activated B cells (NFkB); and d) functional and health-related outcomes, i.e., side-effects and medical outcomes, quality of life (QoL), and functional status.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically confirmed prostate cancer
* Elects prostatectomy as first line treatment (i.e., no androgen ablation, radiation therapy, etc)
* Has at least 3.5 weeks lag-time until scheduled prostatectomy (must be able to participate in the diet and exercise program a full 3.5 weeks).
* Body mass index (BMI) 25 - 49.9
* Mentally competent
* Able to speak and write English
* Has telephone access
* Agrees to be randomized to either study arm (immediate or delayed diet and exercise program)

Exclusion Criteria:

* Another active malignancy (not including non-melanoma skin cancer)
* Medical conditions that affect weight (e.g., untreated thyroid disturbances
* Currently on a weight loss regimen
* Preexisting medical condition(s) that preclude adherence to unsupervised exercise, e.g., severe orthopedic conditions, scheduled for a hip or knee replacement, bone metastases, paralysis, dementia, untreated stage 3 hypertension, or unstable angina, heart attack, congestive heart failure or conditions that dictated hospitalization or oxygen within 6-mths, etc.

Min Age: 19 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-09; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Tumor Proliferation Rate (Ki-67) | Participants will be followed until their prostatectomy (minimum of 3.5 weeks, up to 24 weeks)
  Changes in tumor proliferation rate (Ki-67) over the presurgical study period (minimum of 3.5 weeks, up to 24 weeks) will be explored and compared between the intervention and wait-list control arms.

SECONDARY OUTCOMES:
Changes in body weight and composition, energy intake and physical activity | Participants will be followed until their prostatectomy (minimum of 3.5 weeks, up to 24 weeks)
  Changes in body composition, energy intake and physical activity over the presurgical study period (minimum of 3.5 weeks, up to 24 weeks) will be explored and compared between the intervention and wait-list control arms.

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Demark-Wahnefried, PhD, RD, Principal Investigator — University of Alabama at Birmingham (UAB)
Locations (1):
- University of Alabama at Birmingham (UAB), Birmingham, Alabama, United States

REFERENCES:
- [Result] Demark-Wahnefried W, Nix JW, Hunter GR, Rais-Bahrami S, Desmond RA, Chacko B, Morrow CD, Azrad M, Fruge AD, Tsuruta Y, Ptacek T, Tully SA, Segal R, Grizzle WE. Erratum to: Feasibility outcomes of a presurgical randomized controlled trial exploring the impact of caloric restriction and increased physical activity versus a wait-list control on tumor characteristics and circulating biomarkers in men electing prostatectomy for prostate cancer. BMC Cancer. 2017 Jan 23;17(1):71. doi: 10.1186/s12885-016-3025-3. No abstract available. PMID 28114897
- [Derived] Smith KS, Fruge AD, van der Pol W, Caston NE, Morrow CD, Demark-Wahnefried W, Carson TL. Gut microbial differences in breast and prostate cancer cases from two randomised controlled trials compared to matched cancer-free controls. Benef Microbes. 2021 Jun 15;12(3):239-248. doi: 10.3920/BM2020.0098. Epub 2021 Apr 1. PMID 33789551
- [Derived] Fruge AD, Dasher JA, Bryan D, Rais-Bahrami S, Demark-Wahnefried W, Hunter GR. Physiological Effort in Submaximal Fitness Tests Predicts Weight Loss in Overweight and Obese Men with Prostate Cancer in a Weight Loss Trial. Int J Cancer Clin Res. 2017;4(2):083. doi: 10.23937/2378-3419/1410083. Epub 2017 Oct 16. PMID 29546247
- [Derived] Fruge AD, Ptacek T, Tsuruta Y, Morrow CD, Azrad M, Desmond RA, Hunter GR, Rais-Bahrami S, Demark-Wahnefried W. Dietary Changes Impact the Gut Microbe Composition in Overweight and Obese Men with Prostate Cancer Undergoing Radical Prostatectomy. J Acad Nutr Diet. 2018 Apr;118(4):714-723.e1. doi: 10.1016/j.jand.2016.10.017. Epub 2016 Dec 15. PMID 27988219
- [Derived] Demark-Wahnefried W, Nix JW, Hunter GR, Rais-Bahrami S, Desmond RA, Chacko B, Morrow CD, Azrad M, Fruge AD, Tsuruta Y, Ptacek T, Tully SA, Segal R, Grizzle WE. Feasibility outcomes of a presurgical randomized controlled trial exploring the impact of caloric restriction and increased physical activity versus a wait-list control on tumor characteristics and circulating biomarkers in men electing prostatectomy for prostate cancer. BMC Cancer. 2016 Feb 5;16:61. doi: 10.1186/s12885-016-2075-x. PMID 26850040